CLINICAL TRIAL: NCT01265329
Title: Methods for Objective Selection of Competent Sperm
Acronym: MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Marcos Meseguer, Embryologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0810-C-051-MM
Record Dates: First submitted 2010-10-08; First posted 2010-12-23 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Sperm Selection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No sperm selection
- Annexine V negative (Experimental): Sperm selection with Annexine V protein
  Interventions: Other: Negative selection

INTERVENTIONS:
Other: Negative selection — Sperm selection to continue the treatment with healthy sperm
  Arms: Annexine V negative

SUMMARY:
In spite of the achievements and developement of the assisted reproduction techniques in the last years, there is still an elevated percentage of unsuccessful treatments, needing sometimes repeated attempts to reach pregnancy.

The molecular physiology of sperm is being better characterized, and some reports have demonstrated the implication of different molecular processes in the pathophysiology of male infertility.

Recently, different sperm selection methods have been based on these molecular differences, showing a better quality of the sperm population after selection.

The main objective of this research project is to clinically apply these techniques in order to increase the pregnancy rates per cycle in infertile couples attending assisted reproduction treatments.

ELIGIBILITY:
Inclusion Criteria:

MEN:

- >3million sperm after swimming process

WOMEN:

* < 37 YEARS OLD
* NO GYNECOLOGICAL ANOMOLIES
* HORMONAL VALUES WITHIN CLINICAL RANGE

Exclusion Criteria:

* NONE

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gestation | 14 days
  Sperm selection and blood sample confirming gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Garrido, PhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain